CLINICAL TRIAL: NCT04373265
Title: A Phase 1b, Open-Label Study of Relacorilant in Combination With Pembrolizumab for Patients With Adrenocortical Carcinoma With Excess Glucocorticoid Production
Brief Title: Study of Relacorilant in Combination With Pembrolizumab for Patients With Adrenocortical Carcinoma Which Produces Too Much Stress Hormone (Cortisol)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-551
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; Adrenal Carcinoma; Adrenal Autonomy; Excess Glucocorticoid; Hypertension; Hyperglycemia; Type 2 Diabetes; Impaired Glucose Tolerance; Cortisol; Cushing; Cushing syndrome; Hypercortisolemia; Cushingoid; Moon Face; Dorsocervical Fat Pad; Pembrolizumab; Glucocorticoid Receptor; Relacorilant; GR Antagonist; Adrenal Corticotropic Hormone (ACTH); Adrenocortical Hyperfunction; Adrenal Gland Diseases; Endocrine System Diseases; Pathologic Processes
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Cortex Neoplasms; Hypertension; Hyperglycemia; Diabetes Mellitus, Type 2; Glucose Intolerance; Cushing Syndrome; ACTH Syndrome, Ectopic; Adrenocortical Hyperfunction; Adrenal Gland Diseases; Endocrine System Diseases; Pathologic Processes | interventions — relacorilant; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relacorilant in Combination with Pembrolizumab (Experimental): Participants will be treated on Day -3 to Day 1 (Cohort 1 under fasting conditions) or Day -6 to Day 1 (Cohort 2 under fed conditions) for Cycle 1 only. During the lead-in period, 300 mg relacorilant will be administered daily for 4 -7 days. Patients will receive their first pembrolizumab infusion on Cycle 1 Day 1. The participants will then receive combined treatment from Cycle 1 Day 1 until confirmed PD or unacceptable toxicity. Pembrolizumab will be administered every 6 weeks (on Day 1 of each 42-day cycle) and relacorilant will be administered daily. Optional Cohort 3 will lead-in with 400 mg relacorilant once daily for 7 days and combined treatment of relacorilant and pembrolizumab, depending on PD and toxicity.
  Interventions: Drug: Relacorilant; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Relacorilant — Relacorilant, 100 mg soft gel capsules orally once daily
  Other Names: CORT125134
Drug: Pembrolizumab — Pembrolizumab 400 mg infusion every 6 weeks
  Other Names: Keytruda

SUMMARY:
This study will investigate the safety and efficacy of Relacorilant in combination with Pembrolizumab for Patients with Adrenocortical Carcinoma which Produces Too Much Stress Hormone (Cortisol).

DETAILED DESCRIPTION:
Relacorilant is a small molecule antagonist of the glucocorticoid receptor (GR).

The goal of this study is to assess the safety and efficacy of relacorilant when given in combination with pembrolizumab in patients with advanced adrenocortical carcinoma (ACC) which produces too much stress hormone (cortisol). Too much stress hormone (cortisol) is also called glucocorticoid (GC) excess.

Eligible patients are those with advanced ACC that produces too much cortisol.

Patients will receive treatment until progressive disease (PD) (per RECIST v1.1) is confirmed, experience unmanageable toxicity, or until other treatment discontinuation criteria are met. All patients will be followed for documentation of disease progression, survival information (i.e., date and cause of death) and subsequent treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ACC (advanced unresectable and/or metastatic)
* Measurable disease based upon RECIST v1.1 as determined by the Investigator.
* Documented GC excess (too much cortisol).
* For patients who have received mitotane within 3 months prior to screening, mitotane levels must be <4 mg/L at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Adequate organ and bone marrow function (determined through blood and urine tests)
* Negative pregnancy test for patients of childbearing potential at the Screening and every 6 weeks (+ or - 7 days) in female patients of childbearing potential.

Exclusion Criteria:

* Major surgery within 4 weeks prior to enrollment. If the participant underwent major surgery, they must have recovered adequately prior to starting study treatment.
* Have received and responded (complete response [CR] or partial response [PR]) to prior treatment with any prior checkpoint inhibitor or any other agents targeting T-cell stimulation pathways
* Taking a concomitant medication that is a strong Cytochrome P450 3A (CYP3A) inducer, or that is a substrate of CYP3A with a narrow therapeutic index
* Known untreated parenchymal brain metastasis or have uncontrolled central nervous system (CNS) metastases. Patients must not require steroids and must be neurologically stable without corticosteroids for a minimum of 3 weeks prior to the commencement of the study. Patients with neurologic symptoms must undergo a CT/MRI to rule out occult CNS metastases.
* Requirement for chronic systemic GC treatment, such as active autoimmune disease requiring systemic treatment (corticosteroids or other immunosuppressive medication)
* Patients requiring inhaled glucocorticoids but have no other alternative treatment option if their condition deteriorates during the study.
* Clinically relevant toxicity from prior systemic cytotoxic therapies or radiotherapy that in the opinion of the Investigator has not resolved to NCI-CTCAE v5.0 Grade 1 or less prior to the first dose of relacorilant.
* Treated with the following prior to the first dose of relacorilant:

  1. Any investigational product, systemic anticancer therapy, or radiation therapy within 21 days
  2. Antibodies or anticancer vaccines within 60 days
  3. Mifepristone or other GR antagonists within 5 half-lives of these medications
  4. Adrenostatic medications within 5 half-lives of these medications
* History of severe hypersensitivity to another monoclonal antibody
* Other concurrent cancer or a history of another invasive malignancy within the last 3 years that has a likelihood of recurrence of >30% within the next 5 years. Adequately treated basal and squamous skin cancers, ductal carcinoma in situ, cervical cancer, prostate cancer, non-muscle invasive urothelial cancer or other tumors curatively treated with no evidence of disease are permissible.
* Human immunodeficiency virus (HIV) or current chronic/active infection with hepatitis C virus or hepatitis B virus including: Chronic or active hepatitis B as diagnosed by serologic tests. In equivocal cases, hepatitis B or C polymerase chain reaction may be performed and must be negative for enrollment.
* Clinically significant uncontrolled condition(s) or a condition which, in the opinion of the Investigator, may confound the results of the trial or interfere with the patient's participation, including but not limited to:

  1. Unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction 3 months before study entry.
  2. Active infection that requires parenteral antibiotics.
  3. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | Up to 12 weeks
  Evaluate the percentage of patients with a dose-limiting toxicity

SECONDARY OUTCOMES:
Non-Progression Rate (NPR) | 24 weeks from enrollment
  Evaluate the non-progression rate (NPR) per RECIST v1.1
Progression-Free Survival (PFS) | From date of first treatment, until the date of first documented progression or date of death from any cause, whichever came first, up to month 24
  Evaluate progression-free survival (PFS) per RECIST v1.1
Number of Participants with Adverse Events | Up to 37 days post-treatment
  Adverse events (AEs) by severity grade using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0)
Plasma Concentrations of Relacorilant in Combination with Pembrolizumab in Patients with Advanced ACC and Glucocorticoid Excess | Up to 24 months
  Plasma concentrations of relacorilant in combination with pembrolizumab will be calculated in patients with advanced ACC and glucocorticoid excess

CONTACTS AND LOCATIONS:
Overall Officials: Andreas G Moraitis, MD, Study Director — Corcept Therapeutics
Locations (6):
- United States (6):
  - Site #150, Stanford Cancer Center, Stanford, California
  - Site #007, Moffitt Cancer Center, Tampa, Florida
  - Site #074, University of Michigan Medical School, Ann Arbor, Michigan
  - Site #030 Mayo Clinic, Rochester, Minnesota
  - Site #051, Memorial Hospital, New York, New York
  - Site #183, The University of Texas M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No